CLINICAL TRIAL: NCT04006782
Title: Narrow Dental Implants in Multiple Fixed Prosthesis
Brief Title: Narrow Dental Implants in Multiple Fixed Prosthesis: A Controlled Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIBEA_02_EC_19_Estrechos
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Edentulous Alveolar Ridge
Keywords: edentulous; narrow alveolar ridges
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Narrow dental implants in multiple fixed prosthesis (Other)
  Interventions: Device: Narrow dental implants

INTERVENTIONS:
Device: Narrow dental implants — Insertion of narrow dental implants in multiple fixed prosthesis

SUMMARY:
The objective of this study is to evaluate the survival of narrow dental implants (≤ 3,5 mm) in multiple fixed prostheses in comparison with standard diameter dental implants (≥ 3,75 mm) after 5 years of follow-up. The hypothesis of the study is that narrow dental implants under the evaluated conditions, have the same survival rate and clinical performance than the standard diameter implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (>18 years) of both sexes.
* Clinical need of multiple fixed alveolar ridge rehabilitations.
* Clinical suitability to insert, at least, one narrow dental implant splinted to a standard diameter dental implant.
* Signature of the informed consent

Exclusion Criteria:

* Presence of an active infection
* Being under active treatment with, or have received in the las 30 days treatment with radiotherapy, chemotherapy, immunosuppressors, systemic corticosteroids and/or anticoagulants.
* Presence of severe haematologic disorders.
* Chronic treatment with non steroidal anti-inflammatory drugs (NSAID) or other aniinflammatory drugs.
* Previous diagnosis of chronic hepatitis or liver cirrhosis.
* Presence of Diabetes mellitus with improper metabolic control (glycosylated haemoglobine higher that 9%).
* Patients subjected to dialysis.
* Presence of malignant tumours, haemangioma or angioma in the surgical area.
* History of ischaemic cardiopathy in the las year.
* Pregnancy or plan to getting pregnant during the study.
* Metabolic bone disease
* Patientd receiving treatment with oral or intravenous biphosphonates.
* Any other condition incompatible with the participation in the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Survival after 5 years of follow-up | 5 years in comparison with the baseline
  Implant survival after 5 years of follow-up

SECONDARY OUTCOMES:
Marginal Bone Loss | 1, 3 and 5 years in comparison with the baseline
  Evolution of the peri-implant bone level along the study follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Dental Eduardo Anitua, Vitoria-Gasteiz, Spain

IPD SHARING:
Plan to Share IPD: No